CLINICAL TRIAL: NCT03364894
Title: The Personalized Parkinson Project (De Parkinson Op Maat Studie)
Brief Title: The Personalized Parkinson Project (PPP)
Acronym: PPP
Status: Active, not recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Verily Life Sciences LLC (Industry); University Medical Center Groningen (Other); Maastricht University Medical Center (Other); ParkinsonNet (Unknown); Dutch Parkinson Patient Association (Other); Topsector Life Sciences and Health (Unknown); City of Nijmegen (City Hall) (Unknown); Province of Gelderland (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL59694.091.17
Record Dates: First submitted 2017-11-23; First posted 2017-12-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Biomarkers; Wearable sensors; Imaging; Disease progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen and stool collection from all enrolled patients and cerebrospinal fluid (CSF) from patients who have provided additional and optional consent to CSF collection, for longitudinal genotypic and phenotypic assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background Our understanding of PD has stagnated, partly due to the limited patient diversity and brief followup captured in most study cohorts. Additionally, potentially valuable biomarkers derived from different types of measurements are rarely analyzed in an integrated fashion.

Objective This study aims to create a longitudinal dataset of clinical, molecular, imaging, and continuous wearable sensor-based data from a representative Parkinson's disease (PD) cohort. Data will be made available to researchers worldwide to accelerate the discovery of novel etiological insights, development of new therapeutic approaches, and personalized disease management. For this purpose, an extensible norm for sharing research data will be developed, meeting the latest data privacy and security standards.

Methods Supported by a multinational, public-private partnership, a prospective cohort study was designed to include 650 representative PD patients (disease duration <5 years). Comprehensive follow-up for at least 2 years includes: (1) annual assessment at the study center for acquisition of detailed clinimetric data, magnetic resonance imaging, and biospecimens (plasma, serum, cerebrospinal fluid (CSF), stool) and (2) collection of data from the home environment, using self-assessments and an advanced wrist-worn wearable device to continuously measure biological and environmental signals. Collection, storage, and sharing of these research data will be facilitated by a new method to protect privacy and enhance security using polymorphic encryption and pseudonymization (PEP), a methodology that combines advanced encryption with distributed pseudonymization and data access management.

Conclusion This study is unique, as it includes a cohort of unbiased subjects with recently diagnosed PD, creating an unprecedented dataset that combines longitudinally collected clinical, molecular, imaging, and data from wearable sensors using state of the art technology. The single-center study design minimizes measurement variability. Finally, the innovative methodology for data privacy and protection might serve as a new international standard for sharing research data.

DETAILED DESCRIPTION:
The Personalized Parkinson Project proposes an unbiased approach to biomarker development with multiple clinical, genomic and other molecular, and imaging biomarkers measured in a large population, measured at 3 time points (baseline visit, one year follow-up, and two years' follow-up). In addition, the study protocol includes day-to-day patient monitoring with a multisensor wearable device, the Verily Study Watch, that continuously collects data (movement, pulse, skin temperature, ambient information) and allows for real-time data collection between study visits. The goal of the device is to collect high-resolution, continuous biological signals from the body. These measurements of physiology, activity, and environmental conditions over the course of a 2-year study will be used to create a quantified functional assessment of patients with PD. Mapping these signals with clinical outcomes such as disease progression will allow the investigators to evaluate the relationship between biosensor data and the clinical variables, genotypic, and imaging biomarkers collected in the study.

This study is intended to create a unique resource of genotypic, functional, and phenotypic data collected longitudinally on a cohort of Dutch subjects with PD (n=650), allowing the Research Collaborators to address a series of hypothesis-driven research questions. The aim is to develop novel etiological insights, to identify biomarkers that can assist in predicting differences in prognosis and treatment response between patients, to improve existing treatments, to develop new therapeutic approaches, and to develop a more precise and personalized disease management approach.

Additionally, the cohort will serve as a source of data that can be accessed by qualified researchers worldwide, allowing them to add their research capacity to further address the main aims of this study. For this reason, data governance will be managed by dedicated advisory boards and data review committees, as specified in the study protocol. Participation in this study and results from this study will not be used for patient treatment decisions.

The aim of this study is threefold:

1. The primary objective of the study is to perform a set of hypothesis-driven analyses on the study data set, aiming to correlate established biomarkers (obtained clinically, from brain magnetic resonance imaging (MRI), from cerebrospinal fluid (CSF), from known genetic factors, and from monitoring of biosensors signals) to the rate of disease progression, and to responses to treatment (both pharmacological and behavioral, such as participation in exercise). Also, the investigators aim to identify biomarkers that can assist in predicting differences in prognosis and treatment response between patients. Finally, by developing novel etiological and pathophysiological insights, the study aims to improve existing treatments and to develop new therapeutic approaches, as a basis for development of a more precise and personalized disease management approach.
2. The secondary objective of the study is to evaluate the Verily Study Watch, to assess how these devices could provide information about the function of patients with PD.
3. The tertiary objective of this study is to create an extensive longitudinal dataset describing the genetic, clinical, functional, and phenotypic characteristics of a representative Parkinson's disease (PD) subject cohort (n = 650) to allow researchers to investigate important unanswered questions in PD.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Parkinson's disease of ≤5 years duration, defined as time since diagnosis made by a neurologist.
* Subject is an adult, at least 18 years of age.
* Subject can read and understand Dutch.
* Subject has completed the Informed Consent form, as approved by the Ethics Committee.
* Subject is willing, competent, and able to comply with all aspects of the protocol, including follow-up schedule and biospecimen collection.
* Subject is not a current employee or family member of employees of the institutions involved in the study.

Exclusion Criteria:

* Subject is pregnant or breastfeeding.
* Subject is allergic to nickel.
* Subject has co-morbidities that would hamper interpretation of parkinsonian disability, such as coincident musculoskeletal abnormalities, in the opinion of the Investigator.
* Contraindicated for MRI, e.g. claustrophobia, presence of an active implant, pacemaker, insulin pump, neurostimulator, ossicle prosthesis, and/or other medical device or other non-removable metal part incompatible with MRI.
* For lumbar puncture:

  * Allergy to local anesthetic agents
  * Medical history of compression of spinal cord, current local skin infection at the site of the lumbar puncture, developmental abnormalities in lower spine, blood coagulopathy, anticoagulant medication (Acenocoumarol, Warfarin, Dabigatran).
  * Clinical (or previous MRI) evidence of structural cerebral abnormalities that are not compatible with the performance of a lumbar puncture such as malignancies, abscess, or obstructive hydrocephalus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person with Parkinson's disease who meets the inclusion criteria and does not meet the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Short-term disease progression in terms of motor symptoms | From baseline till 1 year follow-up
  Change in Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III score, measured in off state. This scale assesses 18 motor symptoms (33 items) that are specific for Parkinson's disease. Item scores range from 0 to 4 and are summed, resulting in a total score ranging from 0 to 132, with higher scores representing worse outcomes.
Short-term disease progression in terms of cognitive functioning | From baseline till 1 year follow-up
  Change in Montreal Cognitive Assessment (MoCA) score. The MoCa assesses in 30 items different types of cognitive abilities (0-1 scale), including orientation, short-term memory and attention. All items are summed, resulting in a total score ranging from 0 to 30, with higher scores representing better outcomes.
Mid-term disease progression in terms of motor symptoms | From baseline till 2 year follow-up
  Change in MDS-UPDRS part III score, measured in off state.
Mid-term disease progression in terms of cognitive functioning | From baseline till 2 year follow-up
  Change in Montreal Cognitive Assessment (MoCA) score

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan R Bloem, MD, PhD, Principal Investigator — Radboud university medical center, department of neurology
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The dataset generated in this study will become available to qualified researchers worldwide, provided research questions are approved by the Research and Data Sharing Review Committee (RDSRC). The RDSRC will protect subjects' privacy by limiting the availability of the study data and controlling access to sources of information that might potentially be used to identify the individual subjects associated with the biospecimen analysis.
  The RDSRC will assess the relevance and scientific quality of research proposals for which study data or material is requested. These responsibilities include the consideration of applications for:
  * access to the resources obtained in this study, including data or biomaterials
  * applications for endorsement of a scientific project using study materials;
  * applications for endorsement of a clinical study using study materials.
Supporting Information: Study Protocol
Time Frame: Not decided yet.
Access Criteria: Currently no list of criteria is available.

REFERENCES:
- [Derived] Bloem BR, Marks WJ Jr, Silva de Lima AL, Kuijf ML, van Laar T, Jacobs BPF, Verbeek MM, Helmich RC, van de Warrenburg BP, Evers LJW, intHout J, van de Zande T, Snyder TM, Kapur R, Meinders MJ. The Personalized Parkinson Project: examining disease progression through broad biomarkers in early Parkinson's disease. BMC Neurol. 2019 Jul 17;19(1):160. doi: 10.1186/s12883-019-1394-3. PMID 31315608
- See also: Personalized Parkinson Project study webpage — https://www.parkinsonopmaat.nl/studie